CLINICAL TRIAL: NCT01442766
Title: A Randomised-controlled Trial of Donepezil for Motor Recovery in Acute Stroke
Brief Title: Donepezil Trial for Motor Recovery in Acute Stroke
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No financial support
Sponsor: Imperial College London (Other)
Collaborators: International Stem Cell Forum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO1793
Record Dates: First submitted 2011-09-21; First posted 2011-09-29 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Acute Stroke
Keywords: cholinesterase inhibitor; donepezil; motor; stroke
MeSH Terms: conditions — Stroke | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donepezil (Experimental)
  Interventions: Drug: Donepezil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil — 5mg for 4 weeks, 10mg for 8 weeks if tolerated, or lower dose to continue
  Other Names: Aricept
  Arms: Donepezil
Drug: Placebo — Inert pill that appears identical to donepezil pill. 1 pill for first 4 weeks, followed by 2 pills until end of study.
  Arms: Placebo

SUMMARY:
AIMS: To establish: 1) whether motor deficits in acute stroke improve more in patients taking donepezil, relative to placebo, for 12 weeks; 2) whether brain functional MRI changes as a result of donepezil after 12 weeks.

DETAILED DESCRIPTION:
Stroke is a major personal and social burden, being the commonest cause of severe adult disability. Recovery has been shown in animal models to be dependent upon adequate levels of acetylcholine within the brain - which in stroke is likely to be deficient. This is because acetylcholine-producing nerve cells in the brain are often damaged by strokes.

Consequently, the investigators hypothesise that recovery may be improved by boosting acetylcholine levels in the brain - that can be readily achieved by treating with donepezil.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with acute stroke diagnosed on clinical and neuroimaging grounds who can enter the trial within the 1st week of stroke onset, and who have new motor dysfunction of an upper limb. Motor impairment should be moderate - severe (UE-FM Score ≤50 out of a total of 66).
2. Age: above 18 years old.
3. Patients able and willing to partake in motor tests, and to return for follow-up visit at 12 weeks.
4. Able to understand English.

Exclusion Criteria:

1. Contraindications for donepezil: pregnancy (* Female patients <50 years old will be asked if there is any possibility that they might be pregnant. If there is any uncertainty, or a likelihood that they are pregnant, this will qualify as an exclusion criterion)*; moderate - severe asthma (i.e. regular treatment prescribed for this); bradycardia, syncope, 2nd or 3rd degree heart block, acute or decompensated heart failure; peptic ulcer diagnosed endoscopically and on treatment for this; epilepsy; Parkinson's disease; end-stage renal failure or creatinine > 300 micromol/l; genitourinary tract or gastrointestinal tract obstruction; gastrointestinal tract hemorrhage; myasthenia gravis
2. Other: functionally-significant cognitive impairment (i.e. dementia); significant receptive aphasia (i.e. such that cannot understand purpose or details of trial, and will be unable to cooperate with task instructions); significant physical infirmity as judged by treating physician (e.g. severe organ failure; terminal cancer).
3. Contraindications for MRI (this only pertains for the subset of patients entering the MRI substudy, but is not a contra-indication to the main study providing a diagnosis of stroke is clear from CT): phobia, metal implants including pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11 (Estimated); Primary Completion 2013-11 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Change in Upper Extremity Fugl-Meyer Motor Score (out of 66) over 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Change in Functional MRI Connectivity and Task-related activation (relative % BOLD signal change) over 12 weeks | 12 weeks
  resting-state / activation-related fMRI
Number and type of participants with adverse events | 12 weeks
  Self-reported / Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bentley, MA MRCP PhD, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross Hospital, Imperial College Academic Health Science Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No